CLINICAL TRIAL: NCT00660829
Title: Randomized, Double-Blind, Placebo-Controlled Trial of the Safety and Efficacy of MP03-36 in Subjects With Seasonal Allergic Rhinitis
Brief Title: A Study to Evaluate the Safety and Effectiveness of a Nasal Spray to Treat Seasonal Allergies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP440
Record Dates: First submitted 2008-04-14; First posted 2008-04-17 (Estimated); Results first posted 2010-01-28 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — azelastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Active Comparator): 0.15% Azelastine Hydrochloride
  Interventions: Drug: 0.15% Azelastine Hydrochloride

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: 1
Drug: 0.15% Azelastine Hydrochloride — 0.15% Azelastine Hydrochloride 822 mcg
  Arms: 2

SUMMARY:
The Purpose of this study is to determine if one allergy medication (0.15% azelastine hydrochloride) is more effective than Placebo alone.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients 12 years of age and older with a 2 year history of moderate to severe seasonal allergic rhinitis.
* Must be in generally good health
* Must meet minimum symptom requirements, as specified in the protocol
* Must be willing and able to provide informed consent and to participate in all study procedures
* Positive skin test to a prevalent Texas Mountain Cedar allergen

Exclusion Criteria:

* On Focused Nasal Examination, the presence of any nasal mucosal erosion, nasal ulceration, or nasal septal perforation at either the screening visit or randomization visit will disqualify the subject from the study.
* Other nasal disease(s) likely to affect deposition of intranasal medication, such as sinusitis, rhinitis medicamentosa, clinically significant polyposis, or nasal structural abnormalities.
* Nasal surgery or sinus surgery within the previous year.
* Chronic sinusitis - more than 3 episodes per year
* Planned travel outside of the study area during the study period
* The use of any investigational drug within 30 days prior to Screening. No investigational products are permitted for use during the conduct of this study
* Presence of any hypersensitivity to drugs similar to azelastine and to either sorbitol or sucralose (Splenda® brand sweetener)
* Women who are pregnant or nursing
* Women of childbearing potential who are not abstinent or not practicing a medically acceptable method of contraception
* Respiratory Tract Infections within 14 days prior to screening
* Respiratory Tract Infections requiring antibiotic treatment 14 days prior to screening
* Asthma (with the exception of mild, intermittent asthma). Subjects with mild, intermittent asthma who only require short-acting inhaled bronchodilators (not more often than twice per week) and who do not have nocturnal awakening as a result of asthma are eligible for enrollment
* Significant pulmonary disease including COPD
* Clinically significant arrhythmia or symptomatic cardiac conditions
* A known history of alcohol or drug abuse within the last 2 years
* Existence of any surgical or medical condition or physical or laboratory findings, which in the opinion of the investigator or sponsor's medical monitor, might significantly alter the absorption, distribution, metabolism, or excretion of study drug; that might significantly affect the subject's ability to complete this trial; or their safety in this trial.
* Clinically relevant abnormal physical findings which, in the opinion of the investigator, would interfere with the objectives of the study or that may preclude compliance with the study procedures

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2007-12; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis M Fredane, MD, Study Director — Meda Pharmaceuticals
Locations (6):
- United States (6):
  - Allergy and Asthma Associates, Austin, Texas
  - Allergy and Asthma Center of Austin, Austin, Texas
  - Central Texas Research, New Braunfels, Texas
  - Biogenics Research Institute, San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Allergy and Asthma Center, Waco, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Observation December 13, 2007 Last Observation February 21, 2008
Groups:
- Placebo: Placebo Nasal Spray/2 sprays per nostril once daily for 14 days
- Astepro 0.15%: 0.15% Azelastine Hydrochloride Nasal Spray/2 sprays per nostril once daily for 14 days
Period: Overall Study
Arm/Group | Placebo | Astepro 0.15%
Started | 268 (2 subjects were randomized in error) | 268 (2 subjects were randomized in error)
Completed | 250 | 249
Not Completed | 18 | 19
Not completed — Adverse Event | 3 | 4
Not completed — Lack of Efficacy | 2 | 3
Not completed — Non-Compliance | 0 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 3 | 2
Not completed — Other | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Astepro 0.15% | Total
Number analyzed (Participants) | 266 | 266 | 532
Age, Categorical [Count of Participants; unit: Participants] — Number of participants based on ITT population
  Participants
    <=18 years | 14 | 20 | 34
    Between 18 and 65 years | 241 | 230 | 471
    >=65 years | 11 | 16 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] — Number of participants based on ITT population
  years | 39.5 (14.41) | 40.9 (14.51) | 40.2 (14.46)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of participants based on ITT population
  Participants
    Female | 171 | 175 | 346
    Male | 95 | 91 | 186
Region of Enrollment [Number; unit: participants] — Number of participants based on ITT population
  participants
    United States | 266 | 266 | 532

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 12-hour Reflective Total Nasal Symptom Score (TNSS) (AM and PM Combined)at 14 Days
Description: reflective total nasal symptom score consisting of runny nose, itchy nose, nasal congestion, and sneezing was assessed twice daily. Each symptom is rated on a scale from 0-3: 0=none, 1=mild, 2=moderate, and 3=severe. Total possible score is 24 per day.
  Least Means Square was controlled for study day as the within-patient effect, treatment group and site as the between-patient effects, treatment by-study day interaction, and baseline as co-variate
Time Frame: baseline and 14 days
Population: ITT
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Astepro 0.15%
Number analyzed (Participants) | 266 | 266
Scores on a scale
  Baseline symptom score | 17.98 (3.334) | 18.48 (3.283)
  Overall change from baseline | -1.97 (3.510) | -3.53 (4.241)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.15%; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -1.5633, 95% CI [-2.22 to -0.91], Standard Deviation 0.3345

2. Secondary Outcome: Mean Change From Baseline in Instantaneous Total Nasal Symptom Score (AM) for the Entire 14-day Study Period Compared to Placebo.
Description: End of 24 hour dosing interval: This endpoint is change from baseline in instantaneous (tNSS) for the 14-day study period compared to placebo to observe if the duration of efficacy lasts 24 hours on a day to day basis. Instantaneous (tNSS) consists of runny nose, itchy nose, nasal congestion, and sneezing. Each symptom is rated on a scale from 0-3: 0=none, 1=mild, 2=moderate, and 3=severe.Total possible score is 24 per day.
  Least square means was controlled for study day as the within-patient effect, treatment group and site as the between-patient effects, treatment by-study day interaction, and baseline as a covariate.
Time Frame: baseline and 14 days
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Astepro 0.15%
Number analyzed (Participants) | 266 | 266
Scores on a scale | -0.66 (1.859) | -1.38 (2.103)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.15%; Test type: Superiority or Other; p < 0.001, ANOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -0.7444, 95% CI [-1.07 to -0.42], Standard Error of Mean 0.1677

3. Secondary Outcome: Change From Baseline in 12 Hour Instantaneous Total Nasal Symptom Score (AM and PM Combined) at 14 Days
Description: instantaneous (subjects rate how they feel "right now") total nasal symptom score consisting of runny nose, itchy nose, nasal congestion, and sneezing was assessed twice daily. Each symptom is rated on a scale from 0-3: 0=none, 1=mild, 2=moderate, and 3=severe. Total possible score is 24 per day.
  Least Means Square was controlled for study day as the within-patient effect, treatment group and site as the between-patient effects, treatment by-study day interaction, and baseline as co-variate
Time Frame: baseline and 14-days
Population: ITT
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Astepro 0.15%
Number analyzed (Participants) | 266 | 266
Scores on a scale
  Baseline symptom score | 16.30 (4.054) | 17.06 (4.083)
  Overall change from baseline | -1.52 (3.622) | -2.96 (4.280)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.15%; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -1.4403, 95% CI [-2.11 to -0.77], Standard Deviation 0.3406

4. Secondary Outcome: Change From Baseline in 12-hour Reflective Secondary Symptom Complex Score (SSCS) for the Entire 14-day Study Period Compared to Placebo (AM and PM Combined)
Description: Reflective secondary complex symptom scores (SSCS) (post-nasal drip, itchy eyes, cough and headache) were assessed twice daily. Each symptom is rated on a scale from 0-3: 0=none, 1=mild, 2=moderate, and 3=severe. Total possible SSCS score is 24 per day.
  Least Means Square was controlled for study day as the within-patient effect, treatment group and site as the between-patient effects, treatment by-study day interaction, and baseline as co-variate
Time Frame: baseline and 14-days
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Astepro 0.15%
Number analyzed (Participants) | 266 | 266
Scores on a scale
  Baseline SSCS | 14.40 (4.960) | 14.83 (4.709)
  Change in baseline to Day 14 | -1.52 (3.388) | -2.81 (4.206)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.15%; Change in baseline; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -1.2907, 95% CI [-1.92 to 0.66], Standard Deviation 0.3204

5. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ)
Description: A 28-item RQLQ was completed on Day 1 and Day 14 or Early termination. The RQLQ consists of 7 domains rated on a 7 point scale with 0 being not troubled by the allergy symptoms, and 6 being extremely troubled/all of the time.
  Scores for a series of subscales are not combined for a total overall score, rather domain score will be calculated from the mean score of all items in the domain. Overall score will be calculated from the mean score of all items.
Time Frame: baseline and 14 Days
Population: ITT
Measure: Least Squares Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Astepro 0.15%
Number analyzed (Participants) | 266 | 266
Units on a scale
  Baseline: Overall | 3.68 (1.077) | 3.81 (1.059)
  Change from Baseline:Overall | -0.76 (1.219) | -1.01 (1.304)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.15%; Change from baseline; Test type: Superiority or Other; p = 0.001, ANCOVA

6. Secondary Outcome: Change From Baseline on Direct Visual Nasal Exams at 14 Days
Description: Examination of head and neck (scale: None, Mild, Moderate, Severe) for Epistaxis, Mucosal Edema, Nasal Discharge, Mucosal erythema, Mucosal Bleeding, and Crusting of mucosa. Nasal irritation was rated: 0 = None, Grade 1A = focal irritation, Grade 1B = superficial mucosal erosion, Grade 2 = moderate mucosal erosion, Grade 3 = ulceration, Grade 4 = septal perforation
Time Frame: baseline and 14 Days
Measure: Number; unit: Participants
Arm/Group | Placebo | Astepro 0.15%
Number analyzed (Participants) | 268 | 268
Participants
  Epistaxis: screening - None ( n=268, 268) | 267 | 267
  Epistaxis: screening - Mild ( n=268, 268) | 1 | 1
  Epistaxis: screening - Moderate ( n=268, 268) | 0 | 0
  Epistaxis: screening - Severe ( n=268, 268) | 0 | 0
  Epistaxis: Day 14/ET -None (n=265, 266) | 264 | 265
  Epistaxis: Day 14/ET -Mild (n=265, 266) | 1 | 1
  Epistaxis: Day 14/ET -Moderate (n=265, 266) | 0 | 0
  Epistaxis: Day 14/ET -Severe (n=265, 266) | 0 | 0
  Nasal Irritation: screening - None ( n=268, 268) | 232 | 230
  Nasal Irritation: screening -Grade 1A ( n=268, 268 | 36 | 38
  Nasal Irritation: screening Grade 1B ( n=268, 268) | 0 | 0
  Nasal Irritation: screening -Grade 2 ( n=268, 268) | 0 | 0
  Nasal Irritation: screening -Grade 3 ( n=268, 268) | 0 | 0
  Nasal Irritation: screening -Grade 4 ( n=268, 268) | 0 | 0
  Nasal Irritation: Day 14/ET - none (n=265, 266) | 248 | 251
  Nasal Irritation: Day 14/ET Grade 1A (n=265, 266) | 15 | 15
  Nasal Irritation: Day 14/ET Grade 1B (n=265, 266) | 2 | 0
  Nasal Irritation: Day 14/ET Grade 2 (n=265, 266) | 0 | 0
  Nasal Irritation: Day 14/ET Grade 3 (n=265, 266) | 0 | 0
  Nasal Irritation: Day 14/ET Grade 4 (n=265, 266) | 0 | 0
  Mucosal Edema: screening - none (n= 268, 268) | 18 | 14
  Mucosal Edema: screening - Mild (n= 268, 268) | 55 | 48
  Mucosal Edema: screening - Moderate (n= 268, 268) | 162 | 177
  Mucosal Edema: screening - Severe (n= 268, 268) | 13 | 29
  Mucosal Edema: Day 14/ET none (n=265, 266) | 6 | 17
  Mucosal Edema: Day 14/ET Mild (n=265, 266) | 88 | 77
  Mucosal Edema: Day 14/ET Moderate (n=265, 266) | 152 | 151
  Mucosal Edema: Day 14/ET Severe (n=265, 266) | 19 | 21
  Nasal Discharge: screening - none (n= 268, 268) | 63 | 58
  Nasal Discharge: screening - Mild (n= 268, 268) | 112 | 116
  Nasal Discharge: screening -Moderate (n= 268, 268) | 79 | 82
  Nasal Discharge: screening Severe(n= 268, 268) | 14 | 12
  Nasal Discharge: Day 14/ET none (n=265, 266) | 79 | 72
  Nasal Discharge: Day 14/ET Mild (n=265, 266) | 122 | 128
  Nasal Discharge: Day 14/ET Moderate (n=265, 266) | 64 | 62
  Nasal Discharge: Day 14/ET Severe (n=265, 266) | 0 | 4
  Mucosal Erythema: screening none (n= 268, 268) | 145 | 148
  Mucosal Erythema: screening Mild (n= 268, 268) | 71 | 69
  Mucosal Erythema: screening Moderate (n= 268, 268) | 50 | 48
  Mucosal Erythema: screening Severe (n= 268, 268) | 2 | 3
  Mucosal Erythema: Day 14/ET none (n=265, 266) | 153 | 157
  Mucosal Erythema: Day 14/ET Mild (n=265, 266) | 66 | 63
  Mucosal Erythema: Day 14/ET Moderate (n=265, 266) | 45 | 45
  Mucosal Erythema: Day 14/ET Severe (n=265, 266) | 1 | 1
  Mucosal Bleeding: screening none (n= 268, 268) | 257 | 259
  Mucosal Bleeding: screening Mild (n= 268, 268) | 11 | 8
  Mucosal Bleeding: screening Moderate (n= 268, 268) | 0 | 0
  Mucosal Bleeding: screening Severe (n= 268, 268) | 0 | 0
  Mucosal Bleeding: Day 14/ET none (n=265, 266) | 257 | 256
  Mucosal Bleeding: Day 14/ET Mild (n=265, 266) | 8 | 10
  Mucosal Bleeding: Day 14/ET Moderate(n=265, 266) | 0 | 0
  Mucosal Bleeding: Day 14/ET Severe (n=265, 266) | 0 | 0
  Crusting of Mucosa: screening none (n= 268, 268) | 237 | 245
  Crusting of Mucosa: screening Mild (n= 268, 268) | 25 | 15
  Crusting of Mucosascreening Moderate (n= 268, 268) | 6 | 7
  Crusting of Mucosa: screening Severe (n= 268, 268) | 0 | 1
  Crusting of Mucosa: Day 14/ET - none (n=265, 266) | 245 | 244
  Crusting of Mucosa: Day 14/ET - Mild (n=265, 266) | 14 | 16
  Crusting of Mucosa:Day 14/ET Moderate (n=265, 266) | 6 | 6
  Crusting of Mucosa Day 14/ET Severe( n=265, 266) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Astepro 0.15%
Serious Adverse Events (participants affected / at risk) | 0/266 | 0/266
Other Adverse Events (participants affected / at risk) | 6/266 | 29/266
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=266) | Astepro 0.15% (N=266)
Dysgesusia (Nervous system disorders) | 0 (0) | 12 (12)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 12 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multicenter studies, joint publication is required to assure that the initial publication is based on all data from all sites and investigators participating in these studies agree not to present data gathered individually or by subgroup centers before the initial publication unless jointly agreed by all other investigators and the sponsor. authorship will be determined by mutual agreement.